CLINICAL TRIAL: NCT03268694
Title: Investigation of Oscillations Underlying Human Cognitive and Affective Processing Using Intracranial EEG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Competition with other ongoing projects with this population.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17-1301; R21NS094988-01A1 (NIH)
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Working Memory; Emotions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive and Emotion Processing Tasks (Experimental): As a part of the clinical monitoring, intracranial EEG is continuously collected when the participant is at the Epilepsy Monitoring Unit at the UNC Neuroscience Hospital. We will use an FDA approved EEG amplifier/data acquisition system to collect the research data. Computer-based tasks will be presented through a laptop and task related timing information will be transmitted from the laptop to the data acquisition system. Computer-based tasks will include Working Memory task, Reward Learning Task and Facial Emotion Recognition Task
  Interventions: Behavioral: Working Memory Task; Behavioral: Reward Learning Task; Behavioral: Facial Emotion Recognition Task

INTERVENTIONS:
Behavioral: Working Memory Task — Sternberg Task Items, which can be visually presented alphabets, shapes or numbers or sound tones presented through speakers, will be presented to the participant. The participant will need to maintain the presented items in their memory and indicate, when a single probe item is presented, whether the probe item was present in the immediately preceding list by pressing a key on the keyboard.
  N-Back Task Items are presented continuously sequentially and participants are instructed to indicate whether items are repeated n items before by pressing a key on the keyboard. The task is divided into blocks of 0,1,2,3 -back trials based on the 'n'. For example in the 2 - back task, the participant has to indicate if the item presented 2 items before matches the current item. Similar to the previous task, the items can be presented visually or auditorily.
  Other Names: Sternberg Task; N-Back Task
Behavioral: Reward Learning Task — Two abstract visual stimuli are presented on the screen and participant is asked to choose one. Unknown to the participant, each stimulus is associated with distinct probabilities of virtual reward such that one stimulus is associated with net gain while the other is associated with net loss. The participant's goal is to maximize the reward. Once the participant identifies the stimulus associated with net gain, the reward probabilities are reversed. This process is repeated 5 times.
  Other Names: Learning reversal task
Behavioral: Facial Emotion Recognition Task — On a given trial, participants will be presented with images of two faces side-by-side. The faces will either match in terms of emotion category (e.g., 2 anger faces) or not (e.g., an anger face and a fear face). Faces presented together will always be of the same gender but different identities. Participants will be asked to determine whether the two faces presented depict the same emotion category.

SUMMARY:
Purpose: To investigate the electrophysiological correlates of human cognition and affective processing. Participants: Drug-resistant epilepsy patients undergoing epilepsy surgery cortical mapping with continuous electrocorticography (ECoG) with intracranial electrodes. Procedures (methods): Participants will perform computer-based cognitive and affective processing tasks during routine long-term monitoring. Intracranial EEG will be collected during the task

DETAILED DESCRIPTION:
Oscillations in different frequency bands like theta, alpha, beta, gamma and high gamma are thought to underlie processing of cognitive and emotional information. For example, theta (3 - 7 Hz) and alpha (8 - 12 Hz) oscillations are known to underlie working memory as well as attentional processing. Theta oscillations are known to differentiate emotional and neutral stimuli while gamma oscillations (30 - 50 Hz) are known to underlie rapid integration of information. The fact that these oscillations are also disrupted in neuropsychiatric disorders underline the importance of these oscillations.

A lot of our understanding of these oscillations come from non invasive methods in humans like electroencephalography (EEG), magnetoencephalography (MEG) and invasive methods in animal models. However, EEG and MEG measure oscillations that are generated by collective firing of large cortical patches thereby losing spatial resolution. Also activity from deeper structures like amygdala and hippocampus cannot be picked up in these modalities. Animal models often suffer from the poor translation of behavior from animals to humans and vice versa. Intracranial EEG or Electrocorticography (ECoG) helps overcome the drawbacks described above.

Studies using ECoG have become widespread and have been helpful in elucidating the functional roles of different brain regions in cognition and emotion. The investigators aim to utilize these established procedures to study the role of oscillations recorded from different brain regions in cognition and emotion.

Patients with medically refractory epilepsy undergo long-term invasive monitoring for surgical resection planning. Electrodes are implanted subdurally over seizure focus to identify seizure onset zone and patients are often in the epilepsy monitoring unit at the Neuroscience hospital for approximately a week. During this period, intracranial EEG is constantly acquired for clinical investigation. The investigators plan to recruit these patients while they undergo long-term monitoring to leverage the rare access to direct brain recordings and study the role of oscillations in cognitive and affective processing. Patients who provide informed consent to participate in the study will perform computer based cognitive and emotional processing tasks.

ELIGIBILITY:
Inclusion Criteria:

1. History of medically intractable epilepsy
2. Capable of giving informed consent
3. Aged 18 - 80 years, either sex

Exclusion Criteria:

1. Major systemic illness
2. Severe cognitive impairment defined as mini-mental state examination of less than 20
3. Severe psychiatric illness
4. Excessive use of alcohol or other substances

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2018-07-29 (Actual); Study Completion 2018-07-29 (Actual)

PRIMARY OUTCOMES:
Intracranial EEG Spectra Power | Intracranial EEG will be collected simultaneously when the participants perform the task. 1 Hour
  Spectral analysis of electrophysiology data will be performed using multi-taper fft and wavelet transforms. The measures will be compared between different epochs within the tasks to determine what oscillations are modulated by the task. The correlation between the measures described above and the task performance will also be estimated.

SECONDARY OUTCOMES:
Task Performance: Reaction Times | 1 Hour
  For all the tasks described above, the time from when the response is prompted and when the response is obtained is collected as reaction time. Reaction time is measured in milliseconds.
Intracranial EEG Functional Connectivity Analysis | Intracranial EEG will be collected simultaneously when the participants perform the task. 1 Hour
  Functional connectivity between the different electrodes will be measured using phase locking value and Granger causality.

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Frohlich, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Hae Won Shin, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Hsieh LT, Ranganath C. Frontal midline theta oscillations during working memory maintenance and episodic encoding and retrieval. Neuroimage. 2014 Jan 15;85 Pt 2(0 2):721-9. doi: 10.1016/j.neuroimage.2013.08.003. Epub 2013 Aug 8. PMID 23933041
- [Background] Klimesch W. alpha-band oscillations, attention, and controlled access to stored information. Trends Cogn Sci. 2012 Dec;16(12):606-17. doi: 10.1016/j.tics.2012.10.007. Epub 2012 Nov 7. PMID 23141428
- [Background] Sauseng P, Klimesch W, Heise KF, Gruber WR, Holz E, Karim AA, Glennon M, Gerloff C, Birbaumer N, Hummel FC. Brain oscillatory substrates of visual short-term memory capacity. Curr Biol. 2009 Nov 17;19(21):1846-52. doi: 10.1016/j.cub.2009.08.062. PMID 19913428
- [Background] Symons AE, El-Deredy W, Schwartze M, Kotz SA. The Functional Role of Neural Oscillations in Non-Verbal Emotional Communication. Front Hum Neurosci. 2016 May 25;10:239. doi: 10.3389/fnhum.2016.00239. eCollection 2016. PMID 27252638
- [Background] Bonnefond M, Jensen O. Alpha oscillations serve to protect working memory maintenance against anticipated distracters. Curr Biol. 2012 Oct 23;22(20):1969-74. doi: 10.1016/j.cub.2012.08.029. Epub 2012 Oct 4. PMID 23041197
- [Background] Khader PH, Jost K, Ranganath C, Rosler F. Theta and alpha oscillations during working-memory maintenance predict successful long-term memory encoding. Neurosci Lett. 2010 Jan 14;468(3):339-43. doi: 10.1016/j.neulet.2009.11.028. Epub 2009 Nov 14. PMID 19922772
- [Background] Miller EK, Buschman TJ. Cortical circuits for the control of attention. Curr Opin Neurobiol. 2013 Apr;23(2):216-22. doi: 10.1016/j.conb.2012.11.011. Epub 2012 Dec 22. PMID 23265963
- [Background] Bastos AM, Vezoli J, Bosman CA, Schoffelen JM, Oostenveld R, Dowdall JR, De Weerd P, Kennedy H, Fries P. Visual areas exert feedforward and feedback influences through distinct frequency channels. Neuron. 2015 Jan 21;85(2):390-401. doi: 10.1016/j.neuron.2014.12.018. Epub 2014 Dec 31. PMID 25556836
- [Background] Jacobs J, Kahana MJ. Direct brain recordings fuel advances in cognitive electrophysiology. Trends Cogn Sci. 2010 Apr;14(4):162-71. doi: 10.1016/j.tics.2010.01.005. Epub 2010 Feb 25. PMID 20189441
- [Background] Mendez-Bertolo C, Moratti S, Toledano R, Lopez-Sosa F, Martinez-Alvarez R, Mah YH, Vuilleumier P, Gil-Nagel A, Strange BA. A fast pathway for fear in human amygdala. Nat Neurosci. 2016 Aug;19(8):1041-9. doi: 10.1038/nn.4324. Epub 2016 Jun 13. PMID 27294508
- [Background] Huijgen J, Dinkelacker V, Lachat F, Yahia-Cherif L, El Karoui I, Lemarechal JD, Adam C, Hugueville L, George N. Amygdala processing of social cues from faces: an intracrebral EEG study. Soc Cogn Affect Neurosci. 2015 Nov;10(11):1568-76. doi: 10.1093/scan/nsv048. Epub 2015 May 11. PMID 25964498
- [Background] Murray RJ, Brosch T, Sander D. The functional profile of the human amygdala in affective processing: insights from intracranial recordings. Cortex. 2014 Nov;60:10-33. doi: 10.1016/j.cortex.2014.06.010. Epub 2014 Jun 19. PMID 25043736